CLINICAL TRIAL: NCT01850667
Title: Phase II Multicenter Study of Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma: Toxicity and Outcome
Brief Title: Stereotactic Body Radiation Therapy for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Cancer Center Hospital (Other)
Collaborators: Dongnam Institute of Radiological & Medical Sciences (Other); Soonchunhyang University Hospital (Other); Inje University (Other); Inha University Hospital (Other); Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Mi-Sook Kim, Doctor, Korea Cancer Center Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-1201-001-004; KCT0000454 (Registry Identifier: Clinical Research Information Service); K-1201-001-004 (Other: [Registry ID: Clinical Research information Service)
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Stereotactic body radiotherapy; Stereotactic ablative radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic body radiotherapy (Experimental): Stereotactic body radiotherapy for unresectable hepatocellular carcinoma after incomplete trans-arterial chemo-embolization
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Total stereotactic Body radiotherapy (SBRT) doses will be 60 Gy in 3 fractionations. Patients receive 3 fractionations separated by >48 hours.
  At least 700 ml of normal liver (entire liver minus cumulative GTV) should not receive a total dose of > 17 Gy in three fractions. If volume of normal liver does not exceed 700 ml, at least 70% of normal liver should not receive a total dose of > 17 Gy. In patients without gastroduodenal ulcer on Esophagogastroduodenoscopy (EGD) before SBRT, D2ml of gastrointestinal tract should not exceed 35 Gy. In patients with gastroduodenal ulcer on EGD before SBRT, D2ml of gastrointestinal tract should exceed 28 Gy. (D2ml: minimum dose to 2 ml of gastrointestinal tract)
  Other Names: Stereotactic ablative radiotherapy

SUMMARY:
The standard treatment for hepatocellular carcinoma (HCC) is surgery, such as, by hepatic resection or liver transplantation, but less than 20% of HCC patients are suitable for surgery. In the remaining patients with inoperable and advanced HCC, trans-arterial chemo-embolization (TACE) has been widely used but TACE alone rarely produces complete response and commonly develops recurrence. Recently several small studies reported high tumor response and local control rate after stereotactic body radiotherapy (SBRT) alone or with TACE for inoperable HCC. A single institution phase II trial with SBRT for inoperable HCC after incomplete TACE at Korea Cancer Center Hospital showed promising results: the overall response rate of 73% and 2-year local control rate of 95%. They reported severe gastrointestinal toxicity of 11% because there was no normal tissue constraint for gastrointestinal tract and dosage to gastrointestinal tract was restricted to the lowest levels possible. In addition, they found that the presence of gastroduodenal ulcer before SBRT was significantly influenced on severe gastrointestinal toxicity. Based on this study, we will conduct a multicenter phase II trial on maintenance of treatment results and reduction of severe treatment related toxicity below 5%. To achieve this, we strictly apply normal tissue constraints. Secondly, we will do Esophagogastroduodenoscopy (EGD) before SBRT to evaluate gastroduodenal ulcer. After then, we will apply the normal tissue constraint of gastrointestinal tract according to gastroduodenal ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 20 years of age
* Initially diagnosed or recurrent hepatocellular carcinoma (HCC)
* Unresectable HCC
* Inaccessible to local ablative treatment
* Cirrhotic status of Child Pugh class A or B7
* Eastern Cooperative Oncology Group performance status 0 or 1
* Tumor size < 10cm
* The volume of uninvolved must be at least 700 ml
* Incomplete response after trans-arterial chemo-embolization of 1-5
* A single lesion or multiple lesions including portal vein tumor thrombosis included in radiation field with one or consecutive sessions of SBRT
* No evidence of an uncontrolled lesion at any other site
* No evidence of complications of liver cirrhosis
* No evidence of uncontrolled inter-current illness
* Patient or guardian must be able to provide verbal and written informed consent

Exclusion Criteria:

* Patient with previous history of abdominal radiation
* Direct invasion to esophagus, stomach or colon by HCC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Treatment related toxicity-free survival | 1 year
  From the date of SBRT to the date of treatment related toxicity or last follow-up; Treatment related toxicity will be evaluated by the following criteria.
  1. Adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0;
  2. Classic radiation induced liver disease;
  3. Non-classic Classic radiation induced liver disease;
  4. Worsening of Child-Turcotte-Pugh score;
  5. Worsening of MELD score

SECONDARY OUTCOMES:
Overall survival | 2 years
  From the date of SBRT to the date of death or last follow-up
Progression free survival | 2 years
  From the date of SBRT to the date of first failure or last follow-up
Intrahepatic recurrence free survival | 2 years
  From the date of SBRT to the date of Intrahepatic recurrence or last follow-up
Patterns of failure | 2 years
  Patterns of failure (local, intrahepatic, or systemic)
Systemic failure free survival | 2 years
  From the date of SBRT to the date of systemin failure or last follow-up
Local control rate | 2 years
  From the date of SBRT to the date of local failure or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Sook Kim, MD, PhD, Principal Investigator — Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences
Locations (7):
- South Korea (7):
  - Inje University Haeundae Paik Hospital, Busan
  - Dongnam Institute of Radiological & Medical Sciences, Busan
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Catholic University Incheon St. Mary's Hospital, Incheon
  - Inha University Hospital, Incheon
  - Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences, Seoul
  - Soon Chun Hyang University Hospital Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided